CLINICAL TRIAL: NCT03709654
Title: A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase 1B Study of the Safety, Short-Term Engraftment and Action of NB01 in Adults With Moderate Acne
Brief Title: A Study of the Safety, Engraftment, and Action of Multi-Dosed NB01 in Adults With Moderate Acne
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Naked Biome, Inc. (Industry)
Collaborators: Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NB01-P1BMA
Record Dates: First submitted 2018-10-09; First posted 2018-10-17 (Actual); Results first posted 2020-08-03 (Actual); Last update posted 2020-08-03 (Actual); Status verified 2020-07

CONDITIONS: Acne Vulgaris
Keywords: acne; pimple; black head; white head; zit; probiotic
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Intervention Model Description: Randomized Double Blind Vehicle Controlled Trial, dual arm with 2:1 treatment to vehicle assignment
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Arm (Experimental): Subjects will undergo 1 week lead-in with BPO followed by 11 weeks of NB01 probiotic applied topically.
  Interventions: Biological: NB01
- Vehicle Control (Placebo Comparator): Subjects will undergo 1 week lead-in with BPO followed by 11 weeks of vehicle applied topically.
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Biological: NB01 — 5-7 day pretreatment of gold standard benzoyl peroxide therapy to kill resident facial bacterial followed by 11 weeks of daily topical application of NB01
  Arms: Treatment Arm
Other: Vehicle Control — 5-7 day pretreatment of gold standard benzoyl peroxide therapy to kill resident facial bacterial followed by 11 weeks of daily topical application of vehicle control
  Arms: Vehicle Control

SUMMARY:
Acne vulgaris is a disease caused my multiple factors including overgrowth of bacteria, clogged pores, excessive sebum production and hormonal changes. Recent literature from the Human Microbiome Project has shown there are bacterial strains specific to healthy and acne disease states (Fitz-Gibbon et al, 2013, Johnson et al, 2016, McDowell et al, 2012, Tomida et al, 2013)

From this data, the investigators hypothesize that by eliminating disease-associated bacterial strains and replacing them with health-associated strains, recurrences or flares of acne may be improved, mitigated, and prevented. Instead of current approaches which focus on eliminating all bacteria from the skin, the investigators aim to deliver healthy bacteria to restore the skin to a healthy state via this replacement therapy.

The investigators aim to test this in a Phase Ib multiple application study evaluating the safety, tolerability, and clinical impact that a multiple applications of NB01 have on adult subjects with moderate acne.

DETAILED DESCRIPTION:
A Multicenter, Randomized, Double-Blind, Vehicle-Controlled Phase 1B Study of the Safety, Short-Term Engraftment and Action of NB01 in Adults With Moderate Acne

Acne vulgaris is a multifactorial disease caused by overgrowth of Propionibacterium acnes (P. acnes), impaction of hair follicles, excessive sebum production and hormonal dysregulation. Recent literature from the Human Microbiome Project has shown there are unique microbial signatures specific to healthy and acne disease states.

From this data, the investigators hypothesize that by eliminating resident disease-associated bacterial strains and replacing them with health-associated strains, recurrences/fares of acne may be improved, mitigated, and prevented. Instead of current approaches which focus on eliminating all bacteria from the skin, the investigators aim to deliver healthy bacteria (NB01) to restore the skin to a healthy state via this replacement therapy.

The investigators aim to test this in a Phase 1B multiple application study evaluating the safety, tolerability, and clinical impact that a multiple, daily, applications of NB01 has on adult subjects with moderate acne. Investigators will be profiling the change in microbiome over the course of therapy to determine if exogenously delivered bacteria can populate the skin (engraftment) and cause a shift in the microbiome safely and subsequently impact acne biomarkers that may correlate with clinical disease.

The investigators intend for this therapy to eventually be used in acne subjects with ages ranging from 13-40, and all disease severities as either monotherapy for mild to mild/moderate acne and as an adjuvant therapy for moderate to severe acne at all body sites, with special attention to facial involvement.

This approach is standard to acne therapy whereby mild disease will be treated with a monotherapy (i.e., topical Benzoyl peroxide [BPO]) and moderate/severe disease will be treated with various combinatory regimens (topical antibiotics, BPO, topical retinoids, oral antibiotics).

Primary Objectives:

1. To determine the safety and tolerability of a multiple application of topical P. acnes microbiome transplant ("NB01").

Exploratory Objectives:

1. To define engraftment duration of NB01.
2. To evaluate preliminary clinical efficacy using Acne Lesion Counts (total, inflammatory, and non-inflammatory), Investigator Global Assessment (IGA), and subjective improvement of acne based on subject reported outcomes (Acne QoL Questionnaire).
3. To evaluate treatment effects, based on sebum production in a subpopulation from sites 02 and 03.

Approximately 36 total male and female adult subjects combined with moderate, non-cyclical acne will be enrolled into the trial. Approximately twenty four (24) subjects will be randomly assigned treatment and twelve (12) subjects will be randomly assigned to vehicle control.

This is a multiple topical application study of live bacteria for the study of acne in adult subjects. Following a 5-7 day pretreatment of gold standard benzoyl peroxide therapy to kill resident facial bacterial, 11 weeks of daily topical application of NB01 will be evaluated.

Subject participation in the trial will approximately 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has provided written informed consent.
2. Subject is male or non-pregnant female, 18-40 years of age, inclusive at Screening.
3. Subject has moderate facial acne vulgaris
4. Female subject with non-cyclical acne.
5. Women of childbearing potential (WOCBP) willing to use adequate contraception during study participation
6. Male subjects willing to use an acceptable method of contraception during study participation.
7. Subject has the ability to personally apply benzoyl peroxide (BPO) and study drug, as per protocol.

Exclusion Criteria:

1. Subject has active bacterial, viral, or fungal skin infections.
2. Subject has active nodulocystic acne or acne conglobate, acne fulminans, or other forms of acne (e.g., acne mechanica).
3. Subject is currently participating in an investigational drug, device, or biologic study or has used an investigational drug, biologic or device treatment within 30 days prior to first application of the study drug.
4. Subjects with prosthetic heart valves, pacemakers, intravascular catheters, or other foreign or prosthetic devices/implantable devices/hardware.
5. Subject has a history of chronic human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV) infections.
6. Subject has a history of malignancy (with the exception of non-melanoma skin cancer).
7. Subject is immunosuppressed (such as resulting from transplantation, immunosuppressive therapy, active HIV infection/acquired immune deficiency syndrome [AIDS], neutropenia).
8. Subject had a major surgical procedure, open biopsy, or significant traumatic injury within 14 days of initiating study drug (unless the wound has healed), or anticipation of the need for major surgery during the study.
9. Subjects with close contacts (e.g., spouses, children, or members in the same household) that have severe skin barrier defects or are immunocompromised.
10. Female subject is pregnant or lactating or is planning to become pregnant and/or breast feed within the duration of study participation.

Other entry criteria not listed above will be reviewed of each prospective subject by the study staff to confirm eligibility

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Emma Taylor, MD, Study Director — Naked Biome
Locations (3):
- United States (3):
  - 03, San Diego, California
  - 01, Arlington, Texas
  - 02, Austin, Texas

IPD SHARING:
Plan to Share IPD: No
Initially there is no plan to share IPD. This may change later as the clinical plan develops.

REFERENCES:
- [Result] Fitz-Gibbon S, Tomida S, Chiu BH, Nguyen L, Du C, Liu M, Elashoff D, Erfe MC, Loncaric A, Kim J, Modlin RL, Miller JF, Sodergren E, Craft N, Weinstock GM, Li H. Propionibacterium acnes strain populations in the human skin microbiome associated with acne. J Invest Dermatol. 2013 Sep;133(9):2152-60. doi: 10.1038/jid.2013.21. Epub 2013 Jan 21. PMID 23337890
- [Result] Johnson T, Kang D, Barnard E, Li H. Strain-Level Differences in Porphyrin Production and Regulation in Propionibacterium acnes Elucidate Disease Associations. mSphere. 2016 Feb 10;1(1):e00023-15. doi: 10.1128/mSphere.00023-15. eCollection 2016 Jan-Feb. PMID 27303708
- [Result] McDowell A, Barnard E, Nagy I, Gao A, Tomida S, Li H, Eady A, Cove J, Nord CE, Patrick S. An expanded multilocus sequence typing scheme for propionibacterium acnes: investigation of 'pathogenic', 'commensal' and antibiotic resistant strains. PLoS One. 2012;7(7):e41480. doi: 10.1371/journal.pone.0041480. Epub 2012 Jul 30. PMID 22859988
- [Result] Tomida S, Nguyen L, Chiu BH, Liu J, Sodergren E, Weinstock GM, Li H. Pan-genome and comparative genome analyses of propionibacterium acnes reveal its genomic diversity in the healthy and diseased human skin microbiome. mBio. 2013 Apr 30;4(3):e00003-13. doi: 10.1128/mBio.00003-13. PMID 23631911
- See also: DermNet New Zealand. Acne vulgaris: Acne Grading — http://www.dermnetnz.org/topics/acne-vulgaris
- See also: [FDA] Guidance for Industry: Acne Vulgaris: Developing Drugs for Treatment. Draft: September 2005 — http://www.fda.gov/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM071292
- See also: Early Clinical Trials with Live Biotherapeutic FDA Guidance for Industry: Products: Chemistry, Manufacturing, and Control Information — https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/General/UCM292704.pdf
- See also: FDA Guidance for Industry CGMP for Phase 1 Investigational Drugs — https://www.fda.gov/downloads/BiologicsBloodVaccines/GuidanceComplianceRegulatoryInformation/Guidances/General/UCM292704.pdf

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment Arm | Vehicle Control
Started | 23 | 13
Completed | 20 | 11
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Vehicle Control | Total
Number analyzed (Participants) | 23 | 13 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 24.3 (6.19) | 24.6 (4.7) | 24.4 (5.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 8 | 24
  Male | 7 | 5 | 12
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 7 | 17
  Not Hispanic or Latino | 13 | 6 | 19
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 2
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 3 | 0 | 3
  White | 17 | 12 | 29
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 23 | 13 | 36
Investigator's Global Assessment (IGA) Score - Face [Mean (Standard Deviation); unit: Score on scale] — The investigator assessed the participant's inflammatory lesions on the face using the IGA 5-point scale at screening visit and baseline visits.
  The scale ranges from 0 (best): clear, no evidence of papules or pustules to 4 (worst):
  Score on scale
    IGA at Screening | 3 (0) | 3 (0) | 3 (0)
    IGA at Baseline | 3 (0) | 3 (0) | 3 (0)
Skin bacterial genotype [Mean (Standard Deviation); unit: percentage of genotype] — Skin genotype is the percentage of bacterial population containing health-associated genotypes as measured with TaqMan from a skin swabbed sample.
  percentage of genotype
    deoR/Panbac | 21.8 (24.2) | 26.0 (27.4) | 23.3 (25.4)
    Cas5/Panbac | 7.3 (12.8) | 7.8 (13.0) | 7.5 (12.9)
Lesion Count [Mean (Standard Deviation); unit: number of lesions]
  Inflammatory lesions | 29.1 (7.3) | 30.5 (5.6) | 29.6 (6.7)
  Non-Inflammatory lesions | 35.9 (13.5) | 37.4 (12.8) | 36.4 (13.2)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Changes in Local Skin Reactions
Description: Local Skin Reactions (LSRs) including Erythema, edema, erosion/ulceration, scaling/dryness, and scabbing/crusting scored at Baseline (day of first application) and Week 12 (end of treatment) and reported for each visit as: Absent, Mild, Moderate, or Severe.
  The number of participants (and %) with no change or improvement from Baseline to week 12 visit are reported.
  The number of participants (and %) whose score worsened from Baseline to week 12 visit are reported.
Time Frame: Day 0 through day 80
Population: The Safety population included all randomized subjects who received and applied study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 21 | 12
Participants
  Erythema: No Change / Improved | 19 | 11
  Erythema: Worsened | 2 | 1
  Edema: No Change / Improved | 19 | 9
  Edema: Worsened | 2 | 3
  Erosion/Ulceration: No Change / Improved | 20 | 12
  Erosion/Ulceration: Worsened | 1 | 0
  Scaling/Dryness: No Change / Improved | 16 | 11
  Scaling/Dryness: Worsened | 5 | 1
  Scabbing/Crusting: No Change / Improved | 19 | 12
  Scabbing/Crusting: Worsened | 2 | 0
  Itching: No Change / Improved | 15 | 11
  Itching: Worsened | 6 | 1
  Pain: No Change / Improved | 20 | 12
  Pain: Worsened | 1 | 0

2. Primary Outcome: Number of Participants With Successful Follicular Engraftment of NB01
Description: Follicular engraftment sampling used Biore® Strips at Screening and day 80 (several days after end of treatment).
  The number of subjects with "success" at EOT where "success" is defined as a Follicular Biore® sample with "yes" outcome based on recovery of live NB01at day 80.
Time Frame: 12 weeks
Population: The modified intent-to-treat (mITT) population included all randomized subjects who were dispensed the study drug and had at least 1 post-baseline assessment. Subjects were included in the treatment group to which they were randomized, regardless of the treatment received.
  All randomized subjects (N=36) were included in the mITT population.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
Participants | 1 | 0

3. Primary Outcome: Absolute Change in Genotype Markers: Skin Surface Engraftment "Success"
Description: Skin surface engraftment "success" endpoint is deﬁned by a change in genotype (TaqMan) markers compared to Screening; value is percentage of bacterial population containing health-associated genotype. Result is absolute change from screening value.
Time Frame: Day 0 through day 80
Population: modified intent-to-treat (mITT)
Measure: Mean (Standard Deviation); unit: percentage of bacterial population
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
percentage of bacterial population
  Genotype 1 (deoR), 2 weeks | 6.9 (20.32) | 2.5 (14.17)
  Genotype 1 (deoR), 7 weeks | 5.5 (17.63) | 2.9 (16.96)
  Genotype 1 (deoR), 12 weeks | 3.9 (25.27) | 14.9 (36.76)
  Genotype 2 (Cas 5), 2 weeks | 3.7 (8.16) | 4.8 (12.56)
  Genotype 2 (Cas 5), 7 weeks | 6.6 (17.84) | 3.9 (10.42)
  Genotype 2 (Cas 5), 12 weeks | 4.0 (10.32) | 19.6 (38.69)

4. Primary Outcome: Absolute Change From Screening in Acne Lesion Counts
Description: Reporting absolute change in counts.
Time Frame: Day 0 through day 80
Population: modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
lesion count
  Inflammatory Lesion Count: week 2 | -4.3 (4.77) | -4.7 (6.8)
  Inflammatory Lesion Count: week 7: number analyzed (Participants) | 21 | 12
  Inflammatory Lesion Count: week 7 | -8.4 (6.64) | -6.7 (7.32)
  Inflammatory Lesion Count: week 12: number analyzed (Participants) | 20 | 11
  Inflammatory Lesion Count: week 12 | -15.5 (7.84) | -14.5 (9.56)
  Non-Inflammatory Lesion Count: week 2 | -1.9 (8.89) | -3.0 (6.30)
  Non-Inflammatory Lesion Count: week 7: number analyzed (Participants) | 21 | 12
  Non-Inflammatory Lesion Count: week 7 | -8.6 (8.58) | -9.2 (8.52)
  Non-Inflammatory Lesion Count: week 12: number analyzed (Participants) | 20 | 11
  Non-Inflammatory Lesion Count: week 12 | -15 (16.93) | -17.6 (10.66)

5. Primary Outcome: Percent Change From Screening in Acne Lesion Counts
Description: Efficacy endpoint: Percent change from Screening lesion counts at Day 80 (end of treatment)
Time Frame: Day 0 through day 80
Population: modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: percent change from Baseline
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
percent change from Baseline
  Inflammatory Lesion Count: week 2 | -15.8 (18.72) | -14.8 (20.1)
  Inflammatory Lesion Count: week 7: number analyzed (Participants) | 21 | 12
  Inflammatory Lesion Count: week 7 | -28.9 (20.72) | -20.0 (22.41)
  Inflammatory Lesion Count: week 12: number analyzed (Participants) | 20 | 11
  Inflammatory Lesion Count: week 12 | -54.8 (26.29) | -49.2 (27.19)
  Non-Inflammatory Lesion Count: week 2 | -5.8 (23.99) | -6.2 (16.09)
  Non-Inflammatory Lesion Count: week 7: number analyzed (Participants) | 21 | 12
  Non-Inflammatory Lesion Count: week 7 | -25.0 (23.55) | -21.5 (17.93)
  Non-Inflammatory Lesion Count: week 12: number analyzed (Participants) | 20 | 11
  Non-Inflammatory Lesion Count: week 12 | -43.5 (44.96) | -49 (23.84)

6. Primary Outcome: Number of Participants Achieving "Success" on Investigator Global Assessment (IGA)
Description: The investigator assessed the participant's inflammatory lesions on the face using the Investigator Global Assessment (IGA) 5-point scale.
  The scale ranges from 0 (best): clear, no evidence of papules or pustules to 4 (worst): severe, inflammatory lesions are more apparent, many papules/pustules.
  The outcome is the number of subjects in each treatment group achieving "success" at Week 12; "success" defined as an IGA score of "clear (score=0)" or "almost clear (score=1)" and at least a two-point reduction in IGA compared to Baseline.
Time Frame: Day 0 through day 80
Population: modified intent-to-treat (mITT) population
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
Participants
  Success at 2 weeks | 0 | 0
  Success at 7 weeks | 1 | 0
  Success at 12 weeks | 6 | 1

7. Primary Outcome: Change in Acne QoL Questionnaire Score
Description: At each visit, subjects were asked to complete the Acne Quality of Life [QoL] Questionnaire to assess subjective improvement of acne with 7 response choices ranging from extremely to not at all. The total score ranges from 19 to 114; higher scores reflect improved QoL.
  Outcome measure is absolute change in Acne QoL (Total Score) from Baseline to Day 80.
Time Frame: Day 0 through day 80
Population: modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 23 | 13
score on a scale | 9.7 (16.2) | 33.2 (23.65)

8. Primary Outcome: Absolute Change From Screening in Acne Lesion Counts: Outlier Censored
Description: After reviewing the data, one Treatment Arm subject was found to be an extreme outlier and was censored from this ad-hoc analysis.
  Reporting absolute change in counts.
Time Frame: Day 0 through day 80
Population: Ad Hoc Subject 02-005 (outlier) Censored mITT Population
Measure: Mean (Standard Deviation); unit: lesion count
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 22 | 13
lesion count
  Inflammatory Lesion Count: week 2 | -4.2 (4.82) | -4.7 (6.8)
  Inflammatory Lesion Count: week 7: number analyzed (Participants) | 20 | 12
  Inflammatory Lesion Count: week 7 | -8.5 (6.81) | -6.7 (7.32)
  Inflammatory Lesion Count: week 12: number analyzed (Participants) | 19 | 11
  Inflammatory Lesion Count: week 12 | -15.1 (7.79) | -14.5 (9.56)
  Non-Inflammatory Lesion Count: week 2 | -3.6 (2.77) | -3.0 (6.30)
  Non-Inflammatory Lesion Count: week 7: number analyzed (Participants) | 20 | 12
  Non-Inflammatory Lesion Count: week 7 | -9.7 (7.35) | -9.2 (8.52)
  Non-Inflammatory Lesion Count: week 12: number analyzed (Participants) | 19 | 11
  Non-Inflammatory Lesion Count: week 12 | -18 (10.31) | -17.6 (10.66)

9. Primary Outcome: Percent Change From Screening in Acne Lesion Counts: Outlier Censored
Description: Efficacy endpoint: Percent change from Screening lesion counts at Day 80 (end of treatment)
Time Frame: Day 0 through day 80
Population: Ad Hoc Subject 02-005 Censored mITT Population
Measure: Mean (Standard Deviation); unit: percent change from Baseline
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 22 | 13
percent change from Baseline
  Inflammatory Lesion Count: week 2 | -15.2 (18.91) | -14.8 (20.10)
  Inflammatory Lesion Count: week 7: number analyzed (Participants) | 20 | 12
  Inflammatory Lesion Count: week 7 | -29.0 (21.25) | -20.0 (22.41)
  Inflammatory Lesion Count: week 12: number analyzed (Participants) | 19 | 11
  Inflammatory Lesion Count: week 12 | -53.0 (25.72) | -49.2 (27.19)
  Non-Inflammatory Lesion Count: week 2 | -10.5 (8.55) | -6.2 (16.09)
  Non-Inflammatory Lesion Count: week 7: number analyzed (Participants) | 20 | 12
  Non-Inflammatory Lesion Count: week 7 | -27.8 (20.18) | -21.5 (17.93)
  Non-Inflammatory Lesion Count: week 12: number analyzed (Participants) | 19 | 11
  Non-Inflammatory Lesion Count: week 12 | -51.8 (26.42) | -49.0 (23.84)

10. Primary Outcome: Follicular Engraftment
Description: Follicular communities were genotyped for health-associated loci at both Screening and 12-week visits. The percent increase of Cas5 in multiple communities from each subject is reported.
Time Frame: 12 weeks
Population: modified intent-to-treat (mITT) population
Measure: Mean (Standard Deviation); unit: Percent increase Cas5
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 20 | 11
Percent increase Cas5 | 6518.9 (6711.94) | 492 (939.20)

11. Secondary Outcome: Absolute Change in Sebum Production.
Description: Exploratory Endpoint: Absolute change from Baseline to week 12 in sebum production measured at the mid-glabellar region of the forehead using a Sebumeter.
Time Frame: Day 0 through day 80
Population: modified intent-to-treat subpopulation visiting a subset of sites with a Sebumeter.
Measure: Mean (Standard Deviation); unit: μg/cm^2
Arm/Group | Treatment Arm | Vehicle Control
Number analyzed (Participants) | 19 | 9
μg/cm^2 | 26.2 (52.48) | -22.9 (34.47)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Treatment Arm | Vehicle Control
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/13
Other Adverse Events (participants affected / at risk) | 4/23 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Arm (N=23) | Vehicle Control (N=13)
Application site dryness (General disorders) | 2 (2) | 0 (0)
Application site irritation (General disorders) | 1 (1) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-07-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT03709654/Prot_000.pdf
  • Statistical Analysis Plan (2019-08-15): https://cdn.clinicaltrials.gov/large-docs/54/NCT03709654/SAP_001.pdf